CLINICAL TRIAL: NCT02984449
Title: Preventive Heart Rehabilitation in Patients Undergoing Elective Open Heart Surgery to Prevent Complications and to Improve Quality of Life (Heart-ROCQ) - A Prospective Randomized Open Controlled Trial, Blinded End-point (PROBE)
Brief Title: Preventive Heart Rehabilitation to Prevent Complications in Patients Undergoing Elective Open Heart Surgery
Acronym: Heart-ROCQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, M.A. Mariani, Prof. Dr. M.A. Mariani, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METc: 2016/464 UMCG: 201600576
Record Dates: First submitted 2016-11-29; First posted 2016-12-07 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Coronary (Artery); Disease; Aortic Valve Stenosis; Cardiac Surgery
Keywords: cardiac rehabilitation; surgical complications; quality of life; preoperative; cardiac surgery
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis | interventions — Exercise; Physical Fitness; Nutritional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Double blinding (researcher and participants) is not possible because of logistic reasons. However, the primary endpoint is evaluated by an independent end-point committee, blinded for group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre+postoperative Cardiac rehabilitation (Experimental): receive a cardiac rehabilitation program consisting of three phases. 1) A preoperative optimization phase (3x p/wk, 4-6 weeks, before surgery), 2) a postoperative in-patient phase (15 to 18 days in rehabilitation center, weekend at home) and, 3) an outpatient patient clinical rehabilitation phase (2x p/wk, 4 weeks). During each phase, patients will visit a physical therapist (group sessions of inspiratory muscle training (IMT), strength training, aerobic cycling and breath, cough and relaxation sessions), a dietician and a psychologist to optimize general health and receive advice on lifestyle, anxiety and stress management. Two additional components are coaching to stop smoking
  Interventions: Behavioral: Pre+post-operative Cardiac rehabilitation
- Postoperative Cardiac rehabilitation (Active Comparator): Patients who are randomized to the POST group receive an out-patient cardiac rehabilitation program after surgery. In general, this program starts three to six weeks after discharge (phase ǀǀ) and patients always start with an exercise program, which is supervised by a physical therapist for about six weeks (twice a week). On indication support of psychological and/or dietary consult is added.
  Interventions: Behavioral: Postoperative Cardiac rehabilitation

INTERVENTIONS:
Behavioral: Pre+post-operative Cardiac rehabilitation — CR has the aim to influence favorably the underlying cause of cardiovascular disease, as well as to provide the best possible physical, mental and social conditions (BACPR, 2012).
  Other Names: Exercise; physical fitness; nutrition; psychological support
  Arms: Pre+postoperative Cardiac rehabilitation
Behavioral: Postoperative Cardiac rehabilitation — CR has the aim to influence favorably the underlying cause of cardiovascular disease, as well as to provide the best possible physical, mental and social conditions (BACPR, 2012).
  Other Names: Exercise; physical fitness; nutrition; psychological support
  Arms: Postoperative Cardiac rehabilitation

SUMMARY:
Rationale:

Patients undergoing cardiac surgery are at risk of developing perioperative complications and major adverse cardiac events, mainly related to both their preoperative status and type of surgical procedure. Postoperative exercise based cardiac rehabilitation (CR) is an effective therapy to prolong survival and improve quality of life. However, little is known about the effect on post-operative complications, quality of life and return to work of a combined pre- and post-operative CR program encompassing physical therapy, dietary counseling, psychological support and life style management compared to a CR program, which is provided only after cardiac surgery.

Objective:

to determine whether a pre- and postoperative (PRE+POST) CR program improves the short (up to three months) and long term outcomes (up to one year) of the cardiac surgery (i.e. reduction in postoperative surgical complications, readmissions to hospital and major adverse cardiac events in conjunction with improvements in the physical component of health related quality of life), when compared to postoperative CR only (POST).

Study design:

A Prospective Randomized Open controlled trial, Blinded End-point. Patients are randomized between two standard care CR programs. One group will start a the POST CR program after surgery. The other group will be randomized to a combined PRE+POST CR program.

Study population:

Patients (age > 18 years) admitted for elective coronary bypass surgery, valve surgery and/or aortic surgery

Main study parameters/endpoints:

The primary outcome is a composite weighted endpoint of postoperative surgical complications, re-admissions to hospital, major adverse cardiac events and health related quality of life (two domains: physical functioning and physical problem), at three months and one year after surgery. Endpoints are determined by an independent endpoint committee, blinded to the group allocation. Secondary, the study focuses on physical health (cardiorespiratory fitness, muscle strength and functional status), psychological health (feelings of anxiety and depression), work participation, economics, lifestyle risk factors (physical activity and smoking behavior), self-efficacy and illness representations.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the department of Thoracic Surgery of the UMCG for:
* coronary artery bypass graft surgery
* valve surgery
* aortic surgery
* or a combination of the surgeries mentioned above

Exclusion Criteria:

* Patients accepted for transcatheter aortic valve implantation (TAVI)
* Patients undergoing congenital heart surgery
* Aortic descendens or dissections surgery
* Elite athletes
* Co-morbidities that prevent participation in one or more program elements (e.g. disorders to the nervous or musculoskeletal system that limits exercise capacity, severe COPD (GOLD class 3-4), addiction to alcohol or drugs/ serious psychiatric illness) or when it is undesirable to exercise (e.g. cardiomyopathy/morrow).
* Other treatment planned that possibly will interrupt the program (for example on a waiting list for an organ transplantation, preoperative endocarditis or planned chemotherapy for cancer etc.)
* Unable to read, write and understand Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
a composite weighted score of functional status, postoperative surgical complications, re-admissions to hospital and major adverse cardiac events | Up to one year post-surgery
  Each event, complication or worsening in functional status are considered as a score of 1 to 3 points. These points are summed to calculate the total score.

SECONDARY OUTCOMES:
Atrial fibrillation | up to one year post-surgery
prolonged stay at the intensive care unit | up to one year post-surgery
re-thoracotomy | up to one year post-surgery
re-admissions to intensive care unit | up to one year post-surgery
re-admissions to hospital | up to one year post-surgery
All-cause mortality | up to five year post-surgery
six minutes walking test | Baseline, one day before surgery, 4-7 days, 3-4 months and one year post-surgery
muscle strength | Baseline, one day before surgery, 4-7 days, 3-4 months and one year post-surgery
  This will include grip strength and knee extension
functional status (KATZ) | Baseline, one day before surgery, 4-7 days, 3-4 months and one year post-surgery
Quality of life (Rand-36-v2) | Baseline, one day before surgery, 4-7 days, 3-4 months and one year post-surgery
Depression (PHQ-9) | Baseline, one day before surgery, 4-7 days, 3-4 months and one year post-surgery
Anxiety (GAD) | Baseline, one day before surgery, 4-7 days, 3-4 months and one year after surgery
  Depression (PHQ-9), anxiety (GAD), Quality of life (Rand-36-v2)
iMTA Productivity Cost Questionnaire (PCQ) | Baseline, 3-4, 7-8 and 12 months post-surgery
iMTA Medical Cost Questionnaire (MCQ) | Baseline, 3-4, 7-8 and 12 months post-surgery
Lifestyle risk factors | Baseline, 3-4 months and one year post-surgery
  Physical activity is assessed using the Sensewear GECKO mini-armband (SWA) and the long version (27 questions) of the International Physical Activity Questionnaire (iPAQ)

OTHER OUTCOMES:
Illness perception (IPQ-R), | Baseline, one day before surgery, 4-7 days, 3-4 months and one year post-surgery
Cardiac self-efficacy scale (CSA) | Baseline, one day before surgery, 4-7 days, 3-4 months and one year post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: MA Mariani, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartog J, Blokzijl F, Dijkstra S, DeJongste MJL, Reneman MF, Dieperink W, van der Horst ICC, Fleer J, van der Woude LHV, van der Harst P, Mariani MA. Heart Rehabilitation in patients awaiting Open heart surgery targeting to prevent Complications and to improve Quality of life (Heart-ROCQ): study protocol for a prospective, randomised, open, blinded endpoint (PROBE) trial. BMJ Open. 2019 Sep 18;9(9):e031738. doi: 10.1136/bmjopen-2019-031738. PMID 31537574

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT02984449/Prot_SAP_000.pdf